CLINICAL TRIAL: NCT06225401
Title: Study to Evaluate the Cost-effectiveness of SimCapture for Skills Digital Technology for the Acquisition of Technical Skills Competencies in Peer-to-peer Learning of Undergraduate Nursing Students
Brief Title: Technical Skills Training in Undergraduate Nursing Students: SimCapture for Skills.
Acronym: Simcapture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Barcelona (Other)
Collaborators: Laerdal Medical (Industry)
Responsible Party: Principal Investigator, Marta Raurell-Torreda, Clinical Professor, University of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Simcapture Trial; Facultat Infermeria (Registry Identifier: Universitat de Barcelona)
Record Dates: First submitted 2023-12-31; First posted 2024-01-26 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Education, Nursing Students
Keywords: simulation; deliberate practice; peer to peer learning; technical skills; nursing

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Teacher of nursing students and outcomes assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simcapture PRE (Experimental): In the PRE intervention group (before the traditional teaching) students will practice in pairs, with the same low fidelity simulator, the blood collection technique without a teacher in the classroom. In the SimCapture for Skills interface, the procedure of how to perform the technique (sequence of actions) will be developed in checklist format for the student to check step by step. They will be provided with the same material and classroom time as in traditional teaching (2h).
  Interventions: Other: Simcapture PRE
- Simcapture POST (Experimental): In the POST intervention group (after the traditional teaching) the students will practice in pairs, with the same low fidelity simulator, the blood collection technique without a teacher in the classroom. In the SimCapture for Skills interface, the procedure of how to perform the technique (sequence of actions) will be developed in checklist format for the student to check step by step. They will be provided with the same material and classroom time as in traditional teaching (2h).
  Interventions: Other: Simcapture POST

INTERVENTIONS:
Other: Simcapture PRE — Practice with the SimCapture for Skills interface before the traditional teaching with the teacher in the classroom
  Arms: Simcapture PRE
Other: Simcapture POST — Practice with the SimCapture for Skills interface after the traditional teaching with the teacher in the classroom
  Arms: Simcapture POST

SUMMARY:
Based on the hypothesis that incorporating SimCapture for Skills in the training of technical skills in undergraduate nursing students will increase their competence in the acquisition of technical skills in peer learning, we want to compare the qualification obtained through student self-assessment in the performance of the technique in traditional teaching with classroom teacher versus that obtained with the repetition of the practice with the support of the SimCapture for Skills interface without classroom teacher, as well as the student's perception in terms of satisfaction and self-confidence with both learning spaces. The costs associated with the two types of teaching will also be evaluated.

DETAILED DESCRIPTION:
The traditional teaching with a teacher in the classroom will be received by all the students enrolled in the course. Among these students, two intervention groups will be assigned. One group will train the skills practice with the SimCapture for Skills interface before the traditional teaching with the teacher in the classroom (PRE group) and another group will do it afterwards (POST group).

Skills training:

Prebriefing phase: the court of students, before attending the practice with the low fidelity simulator, both in traditional teaching and teaching with SimCapture, will study in the Virtual Campus of the subject, the procedure of how to perform the technique (sequence of actions) in Word format, and will visualize an example video. They will be administered a knowledge test before the practice to evaluate the acquisition of theoretical concepts.

Simulation phase:

In traditional teaching (2h duration) students will practice in pairs, with the low fidelity simulator, the blood collection technique. The teacher will give them immediate feedback as they practice the technique (zone 0 of the SimZones model). The ratio is 1 teacher to 8 students.

In the PRE intervention group (before the traditional teaching) students will practice in pairs, with the same low fidelity simulator, the blood collection technique without a teacher in the classroom. In the SimCapture for Skills interface, the procedure of how to perform the technique (sequence of actions) will be developed in checklist format for the student to check step by step. They will be provided with the same material and classroom time as in traditional teaching (2h). In each classroom there will be 8 students (4 pairs) and one teacher will supervise 2 classrooms.

In the POST intervention group (after the traditional teaching) the students will practice in pairs, with the same low fidelity simulator, the blood collection technique without a teacher in the classroom. In the SimCapture for Skills interface, the procedure of how to perform the technique (sequence of actions) will be developed in checklist format for the student to check step by step. They will be provided with the same material and classroom time as in traditional teaching (2h). In each classroom there will be 8 students (4 pairs) and one teacher will supervise 2 classrooms.

ELIGIBILITY:
Inclusion Criteria:

* Students enrolled in the compulsory course of the 2nd year of the nursing degree entitled Estades Clíniques I. This subject contains a module called Clinical Skills in which students learn different technical skills with low fidelity simulators (task-trainers).

Exclusion Criteria:

* Not having passed the human anatomy course taught in the 1st year of the nursing degree.
* Not to sign the consent form to participate in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2023-09-13 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2024-04-22 (Actual)

PRIMARY OUTCOMES:
Satisfaction and self-confidence acquired by students in both learning spaces. | Immediately after learning with Simcapture and immediately after learning with the teacher in the classroom
  The Student Satisfaction and Self-Confidence in Learning Scale will be used to evaluate satisfaction and self-confidence, with 12 Likert-rated items (1 -strongly disagree- to 5 -strongly agree-).

SECONDARY OUTCOMES:
Student self-assessment using the technique assessment grid created by the faculty. | During learning with Simcapture or during learning with the teacher in the classroom, through study completion, an average of 3 months
  Checklist technical skills: Rubric with 76 actions to be performed according to the technical procedure. The % of actions correctly performed over the total (n/76*100) will be analyzed.

OTHER OUTCOMES:
Economic costs associated with each type of teaching extrapolating the data to the students enrolled in the subject | Immediately after the learning with Simcapture and with teacher
  Economic costs
Number of times each student can practice the technique with the low-fidelity simulator in both learning spaces. | During learning with Simcapture or during learning with the teacher in the classroom, through study completion, an average of 3 months
  Number of practice for student

CONTACTS AND LOCATIONS:
Overall Officials: Raurell-Torreda Marta, RN, PhD, Principal Investigator — University of Barcelona
Locations (1):
- Faculty of Nursing, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Digital repository
Supporting Information: Study Protocol, ICF
Time Frame: January 2024 to March 2024
Access Criteria: All
URL: https://zenodo.org

REFERENCES:
- See also: Teaching program for intervention groups — https://laerdal.com/es/information/simcapture-for-skills/